CLINICAL TRIAL: NCT00229970
Title: MK0476 Phase II/III Placebo Controlled Double Blind Study
Brief Title: MK0476 Study in Adult Patients With Acute Asthma (0476-322)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-322; MK0476-322; 2005_084
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Experimental): MK0476 7 mg injection
  Interventions: Drug: montelukast sodium
- 3 (Experimental): MK0476 14 mg injection
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — 7 mg or 14 mg single injection
  Arms: 2; 3
Drug: Comparator: Placebo — Placebo single injection
  Arms: 1

SUMMARY:
This study evaluates the efficacy and safety of MK0476 intravenous administration in adult patients with acute asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients With Acute Asthma Attacks

Exclusion Criteria:

* Patient Has Any Known Or Suspected, Acute Or Chronic Cause For Their Pulmonary Symptoms Other Than Asthma (E.G., Copd, Chronic Heart Failure, Etc.)
* Patient Has A Smoking History (20 Cigarettes Per Day) Of More Than 15 Years
* Patient Has A Disease Of The Cardiovascular, Hepatic, Renal, Hematologic Systems, Or Other Severe Disease

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Adachi M, Taniguchi H, Tohda Y, Sano Y, Ishine T, Smugar SS, Hisada S. The efficacy and tolerability of intravenous montelukast in acute asthma exacerbations in Japanese patients. J Asthma. 2012 Aug;49(6):649-56. doi: 10.3109/02770903.2012.690479. Epub 2012 Jun 28. PMID 22742205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III.
  Studied period: September 12, 2005 (date study drug was first administered to first patient) to October 23, 2006 (date study drug was last administered to last patient). Study was conducted at 64 clinical sites.
Pre-assignment Details: Patients with acute exacerbation of bronchial asthma received standard treatments of inhaled β-agonist or oxygen inhalation to treat the acute exacerbations during the 60 minutes in the screening period before the study randomization.
Groups:
- Montelukast 7 mg: Montelukast 7 mg Intravenous Administration
- Montelukast 14 mg: Montelukast 14 mg Intravenous Administration
- Placebo: Placebo Intravenous Administration
Period: Overall Study
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Placebo
Started | 78 | 72 | 75
Completed | 78 | 72 | 75
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Placebo | Total
Number analyzed (Participants) | 78 | 72 | 75 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.5) | 41.5 (13.1) | 42.3 (12.5) | 41.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 34 | 36 | 111
  Male | 37 | 38 | 39 | 114
Asthma Attack Severity based on Asthma Prevention and Management Guideline 2003, Japan [Number; unit: participants] — Mild (Peak Expiratory Flow: 70%-80%), Moderate (Peak Expiratory Flow: 50%-70%), Severe (Peak Expiratory Flow: <=50%) or Serious (Peak Expiratory Flow: incapable measurement, cyanosis, head trip, disturbed consciousness, incontinence or asphyxia)
  participants
    Mild | 54 | 44 | 56 | 154
    Moderate | 23 | 28 | 19 | 70
    Severe | 1 | 0 | 0 | 1
    Serious | 0 | 0 | 0 | 0
Baseline Forced Expiratory Volume in One Second (FEV1) [Mean (Standard Deviation); unit: Liter] | 1.67 (0.55) | 1.62 (0.59) | 1.76 (0.61) | 1.68 (0.58)
Duration of Asthma [Mean (Standard Deviation); unit: Years] | 18.7 (11.5) | 15.46 (11.6) | 17.7 (11.7) | 17.3 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: The Time-weighted Average of Change in Forced Expiratory Volume in One Second (FEV1)
Description: The Time Weighed Average Changes in Forced Expiratory Volume in One Second (FEV1) from pre-allocation baseline over the first 60 minutes after study drug administration with time interval between any measurement and the measurement prior to it is used as the weighting factor
Time Frame: baseline over the first 60 minutes
Population: Last observed value during the 60 minutes treatment period was used in the Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Placebo
Number analyzed (Participants) | 78 | 72 | 75
Liter | 0.09 [0.04 to 0.15] | 0.17 [0.12 to 0.23] | 0.01 [-0.05 to 0.06]
Statistical Analysis 1: Comparison: Montelukast 7 mg vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA; The model included a factor for treatment and using the baseline Forced Expiratory Volume in One Second (FEV1) as a covariate; Mean Difference (Final Values) = 0.09, 95% CI [0.01 to 0.16]
Statistical Analysis 2: Comparison: Montelukast 14 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI [0.09 to 0.24]

ADVERSE EVENTS:
Arm/Group | Montelukast 7 mg | Montelukast 14 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 4 | 4
Other Adverse Events (participants affected / at risk) | 23 | 11 | 13
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Montelukast 7 mg | Montelukast 14 mg | Placebo
Abdominal pain (Gastrointestinal disorders) | 0/78 | 0/72 | 1/75
Acute tonsillitis (Infections and infestations) | 0/78 | 0/72 | 1/75
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/78 | 4/72 | 2/75
Gastritis (Gastrointestinal disorders) | 1/78 | 0/72 | 0/75
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Montelukast 7 mg | Montelukast 14 mg | Placebo
Blood bilirubin increased (Investigations) | 2/77 | 0/72 | 0/75
Blood potassium decreased (Investigations) | 2/76 | 0/72 | 1/73
Blood urine present (Investigations) | 1/75 | 2/70 | 1/75
Bronchitis acute (Infections and infestations) | 0/78 | 2/72 | 0/75
Chest pain (General disorders) | 0/78 | 0/72 | 2/75
Glucose urine present (Investigations) | 4/75 | 0/70 | 1/75
Headache (Nervous system disorders) | 1/78 | 0/72 | 2/75
Nasopharyngitis (Infections and infestations) | 5/78 | 2/72 | 5/75
Protein urine present (Investigations) | 2/75 | 0/70 | 1/75
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4/78 | 1/72 | 0/75
White blood cell count increased (Investigations) | 4/77 | 4/70 | 2/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.